CLINICAL TRIAL: NCT06124521
Title: Increasing Eye Care Utilization in Black Americans At High Risk For Glaucoma Using A Community-Engaged and Faith-Based Intervention
Brief Title: Community Based Treatment for (ComBaT) Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Angela Elam, Assistant Professor of Ophthalmology and Visual Sciences, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00207876; K23MD016430-04 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma
Keywords: Eye Care; Care utilization; Community-based; Faith-based; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye concern (Experimental): Those with a diagnosis of glaucoma or glaucoma suspect (or other concerning eye disease, such as diabetic retinopathy or macular degeneration) will be invited to participate in the ComBaT Glaucoma.
  Interventions: Behavioral: ComBaT Glaucoma

INTERVENTIONS:
Behavioral: ComBaT Glaucoma — ComBaT Glaucoma is a personalized counseling and education program about the participant's diagnosis and the importance of glaucoma follow-up care in maintaining vision.

SUMMARY:
The purpose of this research is to evaluate if intervention and education can change the behavior of someone's willingness to see an eye care provider to prevent blindness and glaucoma. The researchers are investigating if adding additional resources improves participant access to care.

DETAILED DESCRIPTION:
Outcome measures related to acceptability and feasibility are exploratory. They will not be registered or results reported.

ELIGIBILITY:
Inclusion Criteria:

* Black or African American
* Participated in the screening examination portion of the study

Exclusion Criteria:

* Current eye pain (> 8 out of 10)
* Sudden decrease in vision (within 1 week)
* Double vision that doesn't stop when you blink and stops no matter what eye you cover (not blurred, but seeing 2 objects)
* Pregnant women
* Prisoners
* Cognitive impairment- unable to give an ocular and social history
* Moving outside of Michigan or driving distance to the church within 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Eye care utilization | Up to 14 months
  Participants who have not seen an eye care provider for an initial clinical evaluation within 6 months of entering the program or a follow-up evaluation at 12 months will be considered underutilizers. Those who have received evaluation at 6 and 12 months will be considered normal utilizers.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Elam, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Historic King Solomon Baptist Church, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No